CLINICAL TRIAL: NCT02745626
Title: Comparison of Root Resorption, Microbial Colonization & Gingival Health Between Clear Aligners, Self-Ligating Brackets & Conventional Brackets- A Randomized Controlled Clinical Trial
Brief Title: Comparison of Oral Hygiene & Root Resorption During Orthodontic Treatment
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Align Technology, Inc. (Industry)
Responsible Party: Principal Investigator, Madhur Upadhyay, Director (Orthodontic Clinic & Fellowship Program), Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB No. 12-025-2
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Orthodontic Pathological Resorption of External Root; Complication of Personal Oral Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clear Aligner Appliance (Experimental): Clear Aligners, Align Technology Inc., Santa Clara, California
  Interventions: Device: Appliance
- Self-ligating Appliance (Experimental): Carriere Self-Ligating Bracket, Carlsbad, CA
  Interventions: Device: Appliance
- Conventional bracket appliance (Experimental): Preadjusted edge wise brackets using elastomeric ties.
  Interventions: Device: Appliance

INTERVENTIONS:
Device: Appliance — Orthodontic appliance to carry out orthodontic tooth movement.

SUMMARY:
Orthodontic treatment has been traditionally carried out with fixed appliances involving the use of stainless steel brackets and archwires. The challenge has been to move teeth and their roots effectively while minimizing iatrogenic damage such as root resorption and gingival inflammation. In recent years, with the development of new appliances and brackets such as self-ligating brackets and clear aligners there have been reports of improved periodontal status, less iatrogenic root damage and improved hygiene during treatment. Although these treatment modalities have been rapidly accepted in clinical practice, both clinical and basic science research data regarding their overall biological compatibility to support higher levels of evidence based dentistry (e.g, randomized clinical trials) is lacking. In other words, their advantages and disadvantages in this regard have not yet been scientifically evaluated. Such quantification will provide invaluable information for improvements in these treatment modalities.

A randomized controlled clinical trial will be conducted with strict inclusion and exclusion criteria to test the following hypothesis (H) up to 18 months into treatment:

H-1: There is no difference in the amount of root resorption caused by the three different appliances.

H-2: Gingival health is not affected by the 'type of appliance' being used to correct the malocclusion.

H-3: There is no difference in the amount of bacterial count and the type of appliance being used for orthodontic treatment.

The hypothesis will be tested with the following specific aims (SA):

SA-1: To investigate the amount of orthodontically induced inflammatory root resorption generated by treatment.

SA-2: To evaluate the periodontal health of the patients with the different appliance systems.

SA-3: To determine the changes in Streptococcus mutans and total bacterial counts contained in the plaque of orthodontic patients.

SA-4: To ascertain whether there is an association between the microbial count and the type of appliance being used for orthodontic treatment

DETAILED DESCRIPTION:
Importance of the research Orthodontic treatment is no longer limited mainly to children and adolescents. With increasing number of patients from older age groups seeking orthodontic treatment; there has been an increasing demand for esthetic alternatives to conventional fixed stainless steel appliances. Some issues associated with conventional fixed appliances for treatment are: 1) unaesthetic appearance of brackets especially for adult patients, many of whom are unwilling to wear braces, 2) conventional systems compromise the ability of the patient to maintain good oral hygiene; 3) increase the risk of periodontal breakdown due to constant accumulation of plaque around the brackets, wires and ill-fitting bands; 4) require many follow-up visits for appliance reactivation and adjustment if the teeth do not move as desired; 5) iatrogenic root resorption, a major medico-legal concern also poses significant problems for the clinician. Increased use of self-ligating brackets and clear aligners from Invisalign (Align Technology, Inc., Santa Clara, CA) are some of the recent developments in orthodontics that have tried to address these concerns. However clinical evidence highlighting their efficacy has not been quiet forthcoming. Present knowledge is primarily based upon case reports, case series, surveys, anecdotal reports and retrospective studies. In such a scenario it is imperative to find an optimized evidence-based treatment strategy that leads to predictable outcome with complete patient satisfaction during and after treatment while minimizing the risk for root resorption and periodontal breakdown.

RESEARCH DESIGN & METHODS:

Screening procedure:The partcipants were selected from the Division of Orthodontics, Department of Craniofacial Sciences, University of Connecticut, Health Center by two investigators: 1) faculty member supervising the 'clinical component' of the research and 2) faculty member supervising the microbiological and radiological part of the research.

Only after gaining approval from both the faculty members a participant was selected for the study. The participants and their parents were provided with a written explanation on the background of the study, its objectives, and their involvement. In addition to the consent form for routine orthodontic care currently used in the investigator's clinic; the patient or parent/guardian of every participant was given a second consent form specifically related to this study. The following were the inclusion criteria, which were based on previous studies and the investigator's clinical research experience:

1. All the participants should be physically healthy with no relevant allergies or medical problems.
2. All participants ≥ 12 years of age.
3. There should be less than 8mm of anterior crowding or spacing and adequate buccal interdigitation. Patients with posterior edentulous spaces will only be included if treatment does not entail space closure.
4. Participants should have all permanent teeth present, except third molars.
5. Demonstrable ability to maintain adequate oral hygiene.
6. Show optimum dental health without immediate need for restorations.

Following will be the exclusion criteria:

1. Skeletal anterior-posterior discrepancies between the maxilla and mandible (ANB ≥ 5°).
2. Centric relation (CR)- Centric occlusion (CO) discrepancies of greater than 3 mm.
3. Anterior or posterior open bites.
4. Participantswho are pregnant, diabetic or using mouth rinses or interacting medications, including antibiotic therapy.
5. Presence of active periodontal disease.
6. Presence of impacted teeth.
7. Smoking

The participants who fulfilled the above criteria were randomly assigned to one of the treatment groups. The statistician on this project used a computer-generated random numbers ('Rand' function, Microsoft, Excel 2011) for allocation of the sequence. This ensured even distributions of the participants in all the groups. Computer generated random numbers also randomized the right and the left sides of the maxilla for selecting the experimental side.

Sample size From previous studies, it was inferred that a mean colony forming unit (CFU) unit difference of approximately one log (standard deviation (SD) = approximately 1) would result in a clinically significant increase in S.mutans counts. Therefore the sample size of 15 participants per group, at α = 0.05, yielded a statistical power of approximately 0.80 for this study. To account for a 10-25% patient drop out and data loss due to other unavoidable circumstances, we will enroll 68 patients for this study.

Specific aim #1: Measuring the gingival health

Periodontal measurements were recorded specifically for the upper maxillary lateral incisor and second premolar.One individual took all study related periodontal measurements at three different time intervals:

T0: before treatment, T1: after 9 months of treatment &T2: after 18 months of treatment.

During all the measurements, the examiner was blinded from the previous scores. Prior to the start of the research, all participants received standardized oral hygiene instruction to ensure a healthy periodontium.

Goal 1: Measuring the gingival Status The gingival index (GI) developed by Loe and Silness was used.Grades of the severity of gingivitis was scored by clinical inspection based on the size, color, and texture of the gingival margin adjacent to the bracket and bleeding on probing.

Goal 2: Measuring the plaque index (PI) The PI was assessed according to the plaque accumulation in the gingival area in four grades by guiding a probe gingivally over the buccal surface of the selected teeth.

Goal 3: Measuring the papillary bleeding index (PBI) Bleeding on probing (BOP) tendency was measured at the proximal buccal side of the selected teeth, 20 seconds after probing the depth of the pocket/gingival sulcus. The PBI will be assessed in five grades by guiding a probe carefully along the marginal sulcus while observing bleeding intensity.

Specific aim #2: Estimating the total bacterial and Streptococcus mutans count in the plaque sample.

Goal 1: Collection of plaque specimen After isolating the teeth from saliva with cotton rolls and gently drying them to prevent contamination, the supragingival plaque was carefully removed without traumatizing the gingiva, as this would increase the production of gingival crevicular fluid. 52 The plaque-sampling investigator used a standardized protocol to collect specimens at all the three time intervals. Plaque specimens were collected from the labial surfaces immediately surrounding the orthodontic brackets with a sterilized dental scaler with the same tip dimensions (#8/9 Orban DE hoe scaler, Hu-Friedy, Chicago, Ill). Because the area of increased decalcification was generally immediately adjacent to the brackets, four passes, 1 each along the tooth at the bracket interface at the gingival, mesial, distal, and occlusal aspects, were made to avoid overloading the instrument tip. For the invisalign group a single circular stroke around the center of the clinical crown was made. All specimens from each tooth were placed into individual tubes with anonymous coding and sealed for transport to the laboratory. The coding of the specimens ensured blinding of laboratory personnel and help minimize experimental bias.

Goal 2: Microbial sampling Each specimen was diluted in 2 ml of phosphate buffered saline (PBS) dilute yeast extract and the samples will be sonicated for 10 sec before doing serial dilutions. Then 1 ml was submitted to tenfold serial dilution in 9 ml of yeast extract. After each serial dilution the test tubes were vortexed for 10 sec. Ten microlitre (10 μl) of supernatant was then plated onto Tripticase soy agar supplemented with 5% sheep bovine blood (BBL) for total bacterial evaluation and mitis salivarius-bacitracin agar specific for S. mutans. The samples were processed within 2 hours and the plates incubated for 24 hours at 37°C. The number of total CFU (Colony forming unit), specific to S. mutans was identified and counted by the blinded investigator which represented the total recoverable facultative flora.

Specific aim # 3: Estimating the external apical root resorption (EARR) of the maxillary incisors For each patient periapical films of the maxillary incisors and the premolars & orthopantographs (OPG) were taken at the two different time points (T0 & T2). All the periapical films were developed under similar conditions (Dentax 810 Basic) scanned with a ruler to a computer, calibrated and measured in a 1:1 ratio with Adobe Photoshop software (Adobe, San Jose, Calif) for measurement purposes. If required for better interpretation the image of the tooth was enlarged and/or printed.

Measuring root resorption Root and crown length was measured with a sliding caliper to the nearest 0.1 mm The enlargement factor of the second film was adjusted to the first film in each case by reference to the registered crown length, which is assumed to be unchanged by orthodontic treatment.

The 'rule-of-three formula' was applied to calculate root length changes due to orthodontic treatment. It was assumed that during orthodontic treatment the crown length does not change (unless it is fractured). Therefore, the ratio between the initial crown length (C1) and the final crown length (C2) determined the enlargement factor. If no change occured in the root length during treatment, the ratio between the initial root length (R1) and the final root length (R2) should be equal to the C1/C2 ratio. If during treatment the root was shortened, the amount of OIIRR was R1-R2 (C1/ C2).

All research data was identified by unique identifier (Patient1, Patient 2 …) that contained no PHI. Specifically, all data collected from the experiments was not associated with the participant's name, medical ID number, or any other identifier, which could readily identify the participant. All participant data that was gathered was transferred immediately to a secure database where the data was identified only by unique identifiers that were created for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. physically healthy with no relevant allergies or medical problems;
2. above 12 years of age at commencement of treatment;
3. in permanent dentition;
4. less than 5 mm of anterior crowding or spacing with adequate overjet and overbite;
5. ability to maintain adequate oral hygiene
6. in optimum dental health without immediate need for any allied dental procedure.

Exclusion Criteria:

1. skeletal anterior-posterior discrepancies between the maxilla and mandible (ANB ≥ 5°);
2. centric relation - centric occlusion discrepancies of greater than 3 mm;
3. presence of active periodontal disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-12; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Upadhyay, BDS,MDS,MDSc, Principal Investigator — UConn Health
Locations (1):
- Orthodontic Center at University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chhibber A, Agarwal S, Yadav S, Kuo CL, Upadhyay M. Which orthodontic appliance is best for oral hygiene? A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2018 Feb;153(2):175-183. doi: 10.1016/j.ajodo.2017.10.009. PMID 29407494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: December 2011 - March 2014. Location: Orthodontic Clinic, School of Dental Medicine, University of Connecticut Health, Farmington , CT
Period: Overall Study
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Started | 24 | 22 | 22
Completed | 21 | 16 | 19
Not Completed | 3 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance | Total
Number analyzed (Participants) | 21 | 16 | 19 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (4.3) | 14.8 (4.3) | 14.5 (4) | 15.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 9 | 26
  Male | 14 | 6 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 21 | 16 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: A measure of the plaque levels on the desired tooth surface. The following scores were used:
  0 no plaque/debris on inspection and probing
  1. thin film of plaque only visible after probing
  2. ribbon-like layer of plaque covering the sulcus & gingival crown areas but not filling interdental space
  3. thick layer of plaque already visible at inspection and filling interdental space
Time Frame: T0: Before treatment; T1: 9 months of treatment; T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: Plaque Index (PI)
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
Plaque Index (PI)
  T0 (premolar) | 0.5 (0.5) | 0.7 (0.5) | 0.7 (0.5)
  T1(premolar) | 0.8 (0.5) | 1.4 (0.7) | 1.3 (0.7)
  T2(premolar) | 0.9 (0.6) | 1.1 (0.6) | 1.2 (0.7)
  T0(incisor) | 0.6 (0.7) | 0.7 (0.5) | 0.9 (0.9)
  T1 (incisor) | 1 (0.6) | 1.2 (0.5) | 1.5 (1.0)
  T2 (incisor) | 0.9 (0.5) | 1.5 (0.6) | 1.6 (0.8)

2. Secondary Outcome: Gingival Index
Description: An evaluation of the gingival architecture . The following scores were used :
  0 Physiologic gingiva
  1. Mild inflammation (slight color change and little change in texture)
  2. Moderate inflammation (moderate glazing, redness, edema and hypertrophy, bleeding on probing)
  3. Severe inflammation (marked redness and hypertrophy, ulceration. tendency to bleed spontaneously)
Time Frame: T0: Before treatment; T1: 9 months of treatment; T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: Gingival Index (GI)
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
Gingival Index (GI)
  T0 (premolar) | 0.4 (0.5) | 0.1 (0.3) | 0.1 (0.2)
  T1 (premolar) | 0.5 (0.6) | 1 (0.6) | 1.2 (0.8)
  T2 (premolar) | 0.8 (0.5) | 1 (0.7) | 1.1 (0.7)
  T0 (incisor) | 0.6 (0.7) | 0.4 (0.5) | 0.4 (0.6)
  T1 (incisor) | 0.8 (0.7) | 1.2 (0.8) | 1.5 (0.7)
  T2 (incisor) | 1.1 (0.5) | 1.7 (0.7) | 1.5 (0.7)

3. Secondary Outcome: Bleeding Index
Description: An evaluation of the amount of inflammation.
  The following scores were used:
  0 no bleeding
  1. singular bleeding point
  2. several bleeding points or a thin bleeding line along the marginal gingiva
  3. bleeding in the entire interdental gingival triangle immediately after probing
  4. profuse bleeding during probing, bleeding extending over the marginal gingiva eventually with development of blood drops
Time Frame: T0: Before treatment; T1: 9 months of treatment; T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: Bleeding index (BI)
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
Bleeding index (BI)
  T0 (premolar) | 0.5 (0.8) | 0.6 (0.7) | 0.6 (0.7)
  T1 (premolar) | 0.6 (0.8) | 1.4 (1.2) | 1.3 (1.0)
  T2(Premolar) | 0.5 (0.7) | 0.7 (1.1) | 0.8 (0.1)
  T0 (incisor) | 0.7 (0.8) | 0.9 (1) | 0.8 (1)
  T1 (incisor) | 0.5 (0.6) | 1.1 (1) | 1.2 (0.9)
  T2 (incisor) | 0.5 (0.8) | 1.6 (1.2) | 1.3 (1.1)

4. Secondary Outcome: Total Bacterial Count
Description: To calculate the bacterial counts from the diluted plates back to baseline undiluted values, the measurement obtained from the diluted plate was multiplied by 10n (n = number of the serial dilution).
Time Frame: T0: Before treatment; T1: 9 months of treatment; T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: CFU/ml
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
CFU/ml
  T0 | 7.9 (13.8) | 4.7 (15.8) | 4.4 (7.8)
  T1 | 6 (9.9) | 32.7 (92.4) | 10.9 (18.1)
  T2 | 10.6 (14.7) | 9.6 (11.2) | 14.8 (15)

5. Secondary Outcome: S.Mutans Count
Description: as for outcome 4
Time Frame: T0: Before treatment; T1: 9 months of treatment; T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: CFU/ml
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
CFU/ml
  T0 | 0.8 (3.7) | 1 (2.1) | 1.1 (2.1)
  T1 | 0.5 (2) | 0.8 (2.0) | 1.6 (6.5)
  T2 | 0.2 (0.5) | 0.5 (1.2) | 9.9 (1.6)

6. Secondary Outcome: Amount of Root Resorption Observed for Maxillary Lateral Incisor = Length of Root at T0-Length of Root at T2 (in mm)
Description: Root resorption was analyzed by comparing the root length before (T0) treatment and after 18 months of treatment( T2). Therefore the data values indicate the difference in the root length ( in mm).
Time Frame: T0-T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
millimeter (mm) | 0.3 (0.4) | 0.9 (0.9) | 0.8 (1)

7. Secondary Outcome: Amount of Root Resorption Observed for Maxillary Second Premolar = Length of Root at T0-Length of Root at T2 (in mm)
Description: Root resorption was analyzed by comparing the root length before (T0) treatment and after 18 months of treatment( T2)
Time Frame: T0-T2: 18 months of treatment
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Number analyzed (Participants) | 21 | 16 | 19
millimeter (mm) | 0.17 (0.1) | 0.16 (0.11) | 0.21 (0.13)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Clear Aligner Appliance | Self-ligating Appliance | Conventional Bracket Appliance
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
There was no protocol in place to monitor the compliance of the patient with clear aligners.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No